CLINICAL TRIAL: NCT02828085
Title: Improvement of the Etiological Diagnosis of the Pericarditis
Acronym: PERICARDITE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2013-30; 2013-A00962-43 (Other: ANSM)
Record Dates: First submitted 2016-06-30; First posted 2016-07-11 (Estimated); Last update posted 2023-04-21 (Actual); Status verified 2023-04

CONDITIONS: Infective Pericarditis

ARMS (1):
- Infective Pericarditis (Other): In patient prescribed with a pericardite kit for an etiological diagnosis of a pericardial syndrome, an additional nasal swab will be performed in order to perform a specific diagnosis with PCR technique.
  Interventions: Biological: Nasal swab

INTERVENTIONS:
Biological: Nasal swab — Nasal swab will be performed in addition to the routine diagnosis visit in order to determine the diagnosis of infective pericardite with a more specific technique: PCR

SUMMARY:
Pericardial syndrome includes pericardites acute pericardial effusion and cardiac tamponade, recurrent pericarditis squeezing chronic pericarditis. The etiologies are very numerous and can be classified as infectious, neoplastic, metabolic or systemic, toxic causes. Diagnosis is difficult, and 80% of etiologies remain classified idiopathic. In their laboratory to improve the diagnosis of this syndrome investigators have developed a strategy of systematic prescription of biological tests by kit. This prescription by 'kit' strategy proved its interest by comparison with an intuitive requirement of biological. In this study investigators want to improve the diagnostic causative of pericarditis by implementing a new diagnostic strategy. This new strategy includes (i) samples additional less invasive for the patient, the swab pharyngeal and nasal, (ii) the addition of at the outset of more effective diagnostic techniques: specific Polymerase Chain Reaction (PCR)

ELIGIBILITY:
Inclusion Criteria:

* Patient prescribed with a pericarditis kit for etiological diagnosis of a pericardial syndrome.
* Adult patient (= or > 18 years old)
* Patient who freely signed the informed consent form.
* Patient affiliated to a health insurance regime

Exclusion Criteria:

* Minor patient ( age <18 years)
* Pregnant, parturient or breastfeeding woman
* Adult patient incapable or unable to consent
* Patient deprived of liberty under judgment
* Person living in a health or social specialised structure
* Person in vital emergency situation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 979 (Actual)
Dates: Start 2013-07-07 (Actual); Primary Completion 2019-07-24 (Actual); Study Completion 2022-10-26 (Actual)

PRIMARY OUTCOMES:
Percentage of pericarditis whose etiological diagnosis has been established. | 1 day

SECONDARY OUTCOMES:
Identification of the detected emerging pathogens among infectious causesof pericarditis | 1 day
Prevalence of the emerging pathogens: assessement of the percentage of emerging pathogens among the studied population | 1 day

CONTACTS AND LOCATIONS:
Locations (1):
- Assistance Publique Hopitaux de Marseille, Marseille, France